CLINICAL TRIAL: NCT06190704
Title: Prognostic Significance of Coronary Microvascular Dysfunction Assessed by Microvascular Resistance in Hypertrophic Cardiomyopathy Patients
Brief Title: Prognostic Significance of CMD Assessed by IMR in HCM Patients
Acronym: caIMR-HCM
Status: Completed | Type: Observational
Sponsor: Ya-Wei Xu (Other)
Responsible Party: Sponsor-Investigator, Ya-Wei Xu, Chief Physician, Shanghai 10th People's Hospital
Organization: Shanghai 10th People's Hospital (Other)
Other Study IDs: caIMR-HCM
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Coronary Cicrovascular Dysfunction; Hypertrophic Cardiomyopathy Patients
Keywords: Hypertrophic cardiomyopathy; Coronary microvascular dysfunction.; Index of microcirculatory resistance.; Prognosis
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CMD: Microvascular function was assessed using caIMR, and 460 coronary arteries were analyzed. CMD was identified with caIMR>25U, in line with prior research.
  Interventions: Device: caIMR
- non-CMD: Microvascular function was assessed using caIMR, and 460 coronary arteries were analyzed. CMD was identified with caIMR≤25U, in line with prior research.
  Interventions: Device: caIMR

INTERVENTIONS:
Device: caIMR — Coronary angiography-derived IMR (caIMR) is a novel and accurate alternative that can enable the assessment of coronary microvascular function easier, and more efficiently and does not require pressure wire or adenosine.

SUMMARY:
The index of microcirculatory resistance (IMR) serves as an indicator of coronary microvascular dysfunction (CMD) with significant prognostic value in various clinical conditions. However, its impact on CMD in the hypertrophic cardiomyopathy (HCM), whether assessed invasively or non-invasively, is yet to be investigated. We assessed the prognostic importance of CMD using less invasive coronary angiography-derived IMR (caIMR) in HCM patients with nonobstructive epicardial coronary arteries.Patients with HCM who underwent invasive coronary angiography for suspected myocardial ischemia were included. Microvascular function was assessed using caIMR, and 460 coronary arteries were analyzed. CMD was identified with caIMR>25U, in line with prior research, and the primary study endpoint was major adverse cardiac events (MACE).

DETAILED DESCRIPTION:
Patients diagnosed with HCM and referred to the catheterization lab at Shanghai Tenth People's Hospital between 2014 and 2023 for invasive coronary angiography (CAG) due to suspected myocardial ischemia were included in this single-center retrospective observational study. The inclusion criteria of the present study were as follows: 1) Age >18 years old; 2) echocardiographic evidence of HCM, defined as LV myocardial wall thickness of ≥15 mm and or a LV myocardial wall thickness of ≥13 mm in individuals with a family history of HCM, in the absence of an alternative cause for LV hypertrophy. The exclusion criteria were: 1) significant mitral regurgitation; 2) second and third-degree atrioventricular block; 3) presence of significant epicardial coronary stenosis (≥50% stenosis) on CAG; 4) poor life expectancy resulting from concurrent health disease.; and 5) reduced contrast opacification (for caIMR assessment). Our study was conducted in accordance with the Helsinki Declaration and was approved by the ethical review board of Shanghai Tenth People's Hospital.

The essential clinical data, including age, gender, systolic and diastolic blood pressure, heart rate, as well as the past medical history encompassing diabetes, hypertension, hyperlipidemia, stroke, atrial fibrillation, heart failure, family history of HCM, syncope, and smoking history, were systematically recorded. Additionally, laboratory parameters such as total cholesterol, high- and low-density lipoprotein, triglycerides, and N-terminal pro-brain natriuretic peptide were documented. The cardiovascular medical medications, including beta-blockers, antiplatelet agents, ACE inhibitors/ARBs, calcium channel blockers, anticoagulants, diuretics, and amiodarone, for all participants were also noted. Data from electrocardiography, echocardiography, and coronary angiography were diligently collected.

Echocardiography was conducted using an available digital ultrasound system by two cardiologists who were unaware of the clinical data. Measurements, including M mode, standard two-dimensional (2D), and pulsed Doppler, were carried out by the guidelines set by the American Society of Echocardiography. Cardiac dimensions were determined using the average of three cardiac cycles. Parameters such as LV ejection fraction, septal and left posterior wall thickness, left atrium diameter, LV end-systolic diameter, LV end-diastolic diameter, and LV outflow tract gradient were assessed.

Coronary angiography was performed at the operators' discretion, capturing multiple views at either 15 or 30 frames per second. caIMR was determined using the Flash Angio system, consisting of the Flash Angio console, Flash Angio software, and Flash Pressure transducer from Rainmed Ltd., Suzhou, China. A validated protocol utilizing computational pressure-flow dynamics (CPFD) was applied for caIMR estimation in three sequential steps. Initially, a simulated three-dimensional reconstruction of coronary arteries was generated for the targeted vessels. Subsequently, angio-Fractional Flow Reserve (angio-FFR) was estimated using CPFD, incorporating the estimated hyperemic aortic pressure (P'a) based on mean aortic pressure. The calculation of caIMR was then performed using the provided equation:

In this context, (Pd)hyp represents the mean pressure at the distal position during maximal hyperemia, with L denoting a constant representing the length from the inlet to the distal position. The constant K is assigned a value of 2.1, and Vdiastole stands for the mean flow velocity at the distal position during diastole. Additionally, Vhyp is calculated as K multiplied by Vdiastole, signifying the mean flow velocity at the distal position during maximal hyperemia.

caIMR was assessed in at least one of the three coronary arteries for all patients in our study. The epicardial vessel exhibiting the highest caIMR value among the three major coronary vessels was chosen for analysis. In the present study, CMD was identified based on caIMR>25U, consistent with observations from prior research Follow-up was conducted over a mean 43-month period through telephone contact or outpatient visits. The primary clinical endpoints in this study encompassed major adverse cardiac events (MACE), which included: 1) cardiac death: defined as events occurring in the context of cardiac decompensation, pulmonary edema, or progression to end-stage disease, along with other cardiac-related deaths; 2) non-cardiac death: defined as any death occurring during the follow-up period, irrespective of the cause; 3) cardiac readmissions: encompassing hospitalizations for heart failure, myocardial infarction, unstable angina, and malignant arrhythmias; and 4) ischemic stroke: denoting a stroke caused by a blockage in the blood flow to the brain.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old;
* echocardiographic evidence of HCM, defined as LV myocardial wall thickness of ≥15 mm and or a LV myocardial wall thickness of ≥13 mm in individuals with a family history of HCM, in the absence of an alternative cause for LV hypertrophy

Exclusion Criteria:

* significant mitral regurgitation;
* second and third-degree atrioventricular block;
* presence of significant epicardial coronary stenosis (≥50% stenosis) on CAG;
* poor life expectancy resulting from concurrent health disease.;
* reduced contrast opacification (for caIMR assessment)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with HCM and referred to the catheterization lab at Shanghai Tenth People's Hospital between 2014 and 2023 for invasive coronary angiography (CAG) due to suspected myocardial ischemia were included in this single-center retrospective observational study
Sampling Method: Non-Probability Sample
Enrollment: 191 (Actual)
Dates: Start 2014-09-13 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac events (MACE) | Follow-up was conducted over a mean 43-month period through telephone contact or outpatient visits.
  The primary clinical endpoints in this study encompassed major adverse cardiac events (MACE), which included: 1) cardiac death: defined as events occurring in the context of cardiac decompensation, pulmonary edema, or progression to end-stage disease, along with other cardiac-related deaths; 2) non-cardiac death: defined as any death occurring during the follow-up period, irrespective of the cause; 3) cardiac readmissions: encompassing hospitalizations for heart failure, myocardial infarction, unstable angina, and malignant arrhythmias; and 4) ischemic stroke: denoting a stroke caused by a blockage in the blood flow to the brain.

IPD SHARING:
Plan to Share IPD: No